CLINICAL TRIAL: NCT00011583
Title: Robot Assisted Upper Limb Neuro-Rehabilitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Burgar, Charles - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2156
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Acute Stroke
Keywords: Cerebrovascular; Hemiplegia; Robotics
MeSH Terms: conditions — Stroke; Hemiplegia

ARMS (2):
- 1 (Experimental): 1 hour/day of mechanically-assisted upper limb therapy
  Interventions: Device: Robot-assisted therapy
- 2 (Active Comparator): 1 hour/day of upper limb therapy that includes exposure to, but no manipulation by the robot
  Interventions: Device: Traditional therapy

INTERVENTIONS:
Device: Robot-assisted therapy — 1 hour/day of mechanically-assisted upper limb therapy
  Arms: 1
Device: Traditional therapy — 1 hour/day of upper limb therapy that includes exposure to, but no manipulation by the robot
  Arms: 2

SUMMARY:
Our long term objectives are to understand the mechanisms of motor impairment following neurologic injury and to develop interventions to improve motor recovery. A series of complementary, overlapping clinical trials and development activities will validate and optimize the use of robot-assisted upper limb therapy for neuro rehabilitation.

We have developed a robotic system that assists or resists elbow and shoulder movements in three dimensional space. In addition to unilateral exercise modes, a novel bimanual mode enables hemiparetic subjects to practice mirror image upper limb exercises.

DETAILED DESCRIPTION:
Randomized controlled clinical trial of the Mirror Image Movement Enabler (MIME) robotic device for shoulder and elbow neurorehabilitation in subacute stroke patients. MIME incorporates a PUMA 560 robot that applies forces to the paretic limb during unilateral and bilateral movements in three dimensions. Robot-assisted treatment (bilateral, unilateral, and combined bilateral and unilateral) was compared with conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients

Exclusion Criteria:

Unable to follow instructions; medically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2000-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer score | end of training, 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Charles Burgar, MD, Principal Investigator — Central Texas Veterans Health Care System
Locations (1):
- Central Texas Veterans Health Care System, Temple, Texas, United States